CLINICAL TRIAL: NCT05395351
Title: Characteristics and In-hospital Outcomes of Chinese Elderly (>80 Years) Patients With Acute Ischemic Stroke Receiving Intravenous Recombinant Tissue Plasminogen Activator Treatment Within 4.5 Hours of Symptom Onset
Brief Title: Alteplase in Elderly Acute Ischemic Stroke (AIS) Patients During Hospitalization
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0135-0348
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute ischemic stroke (AIS) patients aged >80 years who received IV rt-PA (Alteplase): Group 1: Acute ischemic stroke (AIS) patients aged >80 years who received intravenous recombinant tissue plasminogen activator (IV rt-PA) (Alteplase) within 4.5 hours of symptom onset.
  Interventions: Drug: rt-PA
- Acute ischemic stroke (AIS) patients aged 18 to 80 years who received IV rt-PA (Alteplase): Group 2: Acute ischemic stroke (AIS) patients aged 18 to 80 years who received intravenous recombinant tissue plasminogen activator (IV rt-PA) (Alteplase) within 4.5 hours of symptom onset.
  Interventions: Drug: rt-PA
- Acute ischemic stroke (AIS) patients aged >80 years without thrombolysis treatment: Group 3: Acute ischemic stroke (AIS) patients aged >80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment.
- Acute ischemic stroke (AIS) patients aged 18 to 80 years without thrombolysis treatment: Group 4: Acute ischemic stroke (AIS) patients aged 18 to 80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment.

INTERVENTIONS:
Drug: rt-PA — Intravenous recombinant tissue plasminogen activator (IV rt-PA)
  Other Names: Alteplase
  Groups: Acute ischemic stroke (AIS) patients aged 18 to 80 years who received IV rt-PA (Alteplase); Acute ischemic stroke (AIS) patients aged >80 years who received IV rt-PA (Alteplase)

SUMMARY:
The objective of the study is to find out the in-hospital clinical outcomes among Chinese Acute Ischaemic Stroke (AIS) patients, who were treated with intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) within 4.5 hours of symptom onset in different age groups (18 to 80 years and above 80 years).

ELIGIBILITY:
Inclusion Criteria:

* Patient registered in the Chinese Stroke Centre Alliance (CSCA) platform from Aug 2015 to Jul 2019
* ≥18 years old
* Diagnosed as Acute Ischemic Stroke (AIS) at admission
* Arrived or admitted into hospital within 4.5 hours of symptom onset
* For patients in the iv rt-PA groups only: received IV rt-PA within 4.5 hours of symptom onset

Exclusion Criteria:

* Documented Intravenous Thrombolysis (IVT) absolute contraindication
* Key data missing (age, gender, baseline National Institutes of Health Stroke Scale [NIHSS], time of symptom onset, IVT treated or not, time of IV alteplase treatment)
* Received thrombolysis agents other than IV rt-PA (urokinase, tenecteplase, recombinant plasminogen activator, prourokinase, streptokinase)
* Received endovascular treatment
* Received IV rt-PA after 4.5 hours of symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke (AIS) patients who were treated with Intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) or did not receive thrombolysis treatment within 4.5 hours of symptom onset, aged ≥18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 113035 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim (China) Investment Co., ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Jiang Y, Wang C, Gu H, Zhou Q, Jiang Y, Li Z, Wang Y. In-hospital outcomes of intravenous recombinant tissue plasminogen activator treatment for acute ischemic stroke in patients aged >80 years: Findings from the Chinese Stroke Center Alliance. J Stroke Cerebrovasc Dis. 2025 Jan;34(1):108102. doi: 10.1016/j.jstrokecerebrovasdis.2024.108102. Epub 2024 Oct 28. PMID 39477171
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study the Chinese Stroke Centre Alliance (CSCA) data was used to describe the in-hospital clinical outcomes regarding safety and effectiveness for acute ischemic stroke (AIS) patients who were treated with intravenous recombinant tissue plasminogen activator (IV rt-PA) within 4.5 hours of symptom onset, aged above 80 years, as well as between 18 and 80 years.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Without Thrombolysis Treatment | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Without Thrombolysis Treatment
Started | 3332 | 28086 | 12533 | 69084
Completed | 3332 | 28086 | 12533 | 69084
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Without Thrombolysis Treatment | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Without Thrombolysis Treatment | Total
Number analyzed (Participants) | 3332 | 28086 | 12533 | 69084 | 113035
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.4 (3.2) | 63.2 (10.7) | 84.9 (3.4) | 64.2 (10.4) | 66.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1710 | 9188 | 6418 | 24409 | 41725
  Male | 1622 | 18898 | 6115 | 44675 | 71310
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality During Hospitalization of Acute Ischemic Stroke (AIS) Patients
Description: All-cause mortality during hospitalization of acute ischemic stroke (AIS) patients who received intravenous recombinant tissue plasminogen activator (IV rt-PA).
Time Frame: Up to 100 days.
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission who received intravenous recombinant tissue plasminogen activator (IV rt-PA) (Alteplase). Endpoint was planned to only include Group 1 and 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 3332 | 28086
Percentage of participants | 2.6 [2.1 to 3.2] | 0.8 [0.7 to 0.9]

2. Secondary Outcome: Percentage of Patients With Hemorrhagic Stroke During Hospitalization
Description: Percentage of patients with hemorrhagic stroke during hospitalization.
Time Frame: Up to 100 days.
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission. Endpoint was planned to only include Group 1 and 2.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 3332 | 28086
Percentage of subjects | 6.7 [5.8 to 7.5] | 3.1 [2.9 to 3.3]

3. Secondary Outcome: Change of NIHSS Score From Before Intravenous Recombinant Tissue Plasminogen Activator (IV Rt-PA) Treatment to 24 Hours After IV Rt-PA Treatment
Description: The National Institutes of Health Stroke Scale (NIHSS) is a scale of stroke severity, it ranges from 0 to 42 where a score of 0 indicates no stroke symptoms and higher scores indicate incremental levels of neurologcial impairment.
Time Frame: Up to 24 hours.
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission. Endpoint was planned to only include Group 1 and 2. Only patients with collected NIHSS scores were included in the endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 1404 | 10652
Score on a scale | 2.8 (5.0) | 2.5 (4.3)

4. Secondary Outcome: Modified Rankin Score (mRS) at Discharge
Description: The Modified Rankin Score (mRS) ranges from 0 to 6, where 0 indicates no symptoms, 1 no significant disability, 2 slight disability, 3 moderate disability, 4 moderately severe disability, 5 severe disability and 6 death.
Time Frame: Up to 100 days.
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission. Subjects without a discharge mRS score were excluded. Endpoint was planned to only include Group 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 2325 | 18674
Participants
  mRS score 0 | 383 | 5447
  mRS score 1 | 612 | 6427
  mRS score 2 | 281 | 2131
  mRS score 3 | 216 | 1393
  mRS score 4 | 399 | 2163
  mRS score 5 | 346 | 902
  mRS score 6 | 88 | 211

5. Secondary Outcome: Number of Patients With Stroke Recurrence During Hospitalization
Description: Number of patients with stroke recurrence during hospitalization.
Time Frame: Up to 100 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 3332 | 28086
Participants | 369 | 2039

6. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization.
Time Frame: Up to 100 days.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase)
Number analyzed (Participants) | 3318 | 27952
days | 12.7 (9.6) | 11.5 (7.6)

7. Secondary Outcome: Percentage of Intravenous Recombinant Tissue Plasminogen Activator (IV Rt-PA) Treatment Among Acute Ischemic Stroke (AIS) Patients Arrived or Were Admitted to the Hospital Within 4.5 Hours of Symptom Onset
Description: Percentage of intravenous recombinant tissue plasminogen activator (IV rt-PA) treatment among acute ischemic stroke (AIS) patients arrived or were admitted to the hospital within 4.5 hours of symptom onset.
Time Frame: Up to 4.5 hours.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Acute Ischemic Stroke (AIS) Patients Aged >80 Years: Group 1: Acute ischemic stroke (AIS) patients aged >80 years who received intravenous recombinant tissue plasminogen activator (IV rt-PA) (Alteplase) within 4.5 hours of symptom onset.
  and Group 3: Acute ischemic stroke (AIS) patients aged >80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment.
- Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years: Group 2: Acute ischemic stroke (AIS) patients aged 18 to 80 years who received intravenous recombinant tissue plasminogen activator (IV rt-PA) (Alteplase) within 4.5 hours of symptom onset.
  and Group 4: Acute ischemic stroke (AIS) patients aged 18 to 80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment.
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years
Number analyzed (Participants) | 15865 | 97170
Percentage of participants | 21.0 [20.4 to 21.6] | 28.9 [28.6 to 29.2]

8. Secondary Outcome: Percentage of Intravenous Recombinant Tissue Plasminogen Activator (IV Rt-PA) Treatment Within 4.5 Hours of Symptom Onset Among Eligible AIS Patients (3.5-hour Arrival or Admission)
Description: Percentage of intravenous recombinant tissue plasminogen activator (IV rt-PA) treatment within 4.5 hours of symptom onset among eligible AIS patients (3.5-hour arrival or admission).
Time Frame: Up to 4.5 hours.
Population: Patients registered in the Chinese Stroke Centre Alliance (CSCA) platform from August 2015 to July 2019 with an acute ischemic stroke (AIS) diagnoses at admission and who arrived to the hospital within 3.5 hours of symptom onset and who were eligible for rt-PA treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Acute Ischemic Stroke (AIS) Patients Aged >80 Years: Acute ischemic stroke (AIS) patients aged >80 years who arrived at the hospital within 3.5 hours of symptom onset and were eligible for recombinant tissue plasminogen activator (rt-PA) treatment.
- Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years: Acute ischemic stroke (AIS) patients aged 18 to 80 years who arrived at the hospital within 3.5 hours of symptom onset and were eligible for recombinant tissue plasminogen activator (rt-PA) treatment.
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years
Number analyzed (Participants) | 13639 | 84982
Percentage of participants | 23.9 [23.2 to 24.6] | 32.2 [31.8 to 32.5]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study. All-cause mortality was only collected and reported for group 1 and group 2 for up to 100 days.
Description: This is a non-interventional study using electronic health care records, with data retrieved from the Chinese Stroke Centre Alliance (CSCA). No adverse events were collected on an individual case level. All-cause mortality was only collected and reported for group 1 and group 2.
Arm/Group | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Who Received IV Rt-PA (Alteplase) | Acute Ischemic Stroke (AIS) Patients Aged >80 Years Without Thrombolysis Treatment | Acute Ischemic Stroke (AIS) Patients Aged 18 to 80 Years Without Thrombolysis Treatment
All-Cause Mortality (participants affected / at risk) | 88/3332 | 211/28086 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Hospital participation in the Chinese Stroke Centre Alliance (CSCA) was voluntary. To avoid selection bias, all patients were included without sampling when dataset was extracted. The larger sample size and broad geological distribution increased representativeness.

Data collected by hospitals were not audited by external chart review. Data reliability depends on training for data abstractors and automated checks to identify erroneous, illogical data entries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT05395351/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05395351/SAP_001.pdf